CLINICAL TRIAL: NCT05576623
Title: A Phase I/II (Single Center, Open, Phase I and Multicenter, Double-Blinded, Randomized, Placebo-Controlled, Phase II) Trial to Evaluate the Safety and Immunogenicity of the AdCLD-CoV19-1 OMI Administered as a Booster to Healthy Adults Aged 19 Years Old and Above
Brief Title: Safety and Immunogenicity of AdCLD-CoV19-1 OMI as a Booster: A SARS-CoV-2 (COVID-19) Preventive Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVENT-201
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Vaccines
Keywords: COVID-19; SARS-CoV-2; Omicron; B.1.1.529
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 dose of AdCLD-CoV19-1 OMI (Part A) (Experimental): Group in Part A will receive 1 dose of AdCLD-CoV19-1 OMI
  Interventions: Biological: AdCLD-CoV19-1 OMI (Part A)
- 1 dose of AdCLD-CoV19-1 OMI (Part B) (Experimental): Group 1 in Part B will receive 1 dose of AdCLD-CoV19-1 OMI
  Interventions: Biological: AdCLD-CoV19-1 OMI (Part B)
- Placebo (Part B) (Placebo Comparator): Group 2 in Part B will receive 1 dose of placebo
  Interventions: Other: Placebo (Part B)

INTERVENTIONS:
Biological: AdCLD-CoV19-1 OMI (Part A) — 20 participants will receive investigational product (AdCLD-CoV19-1 OMI) via intramuscular injection in the deltoid muscle
  Arms: 1 dose of AdCLD-CoV19-1 OMI (Part A)
Biological: AdCLD-CoV19-1 OMI (Part B) — 250 participants will receive investigational product (AdCLD-CoV19-1 OMI) via intramuscular injection in the deltoid muscle
  Arms: 1 dose of AdCLD-CoV19-1 OMI (Part B)
Other: Placebo (Part B) — 50 participants will receive placebo via intramuscular injection in the deltoid muscle
  Arms: Placebo (Part B)

SUMMARY:
The safety and immunogenicity of AdCLD-CoV19-1 OMI (5.0x10^10 VP (0.5 mL)/dose/Vial) administered as a booster in healthy adults aged 19 years old and above will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. (Part A) Individual aged between 19-64 years old and willing to provide written informed consent to participate study voluntarily.

   (Part B) Individual aged 19 years and above and willing to provide written informed consent to participate study voluntarily.
2. Individual fall under one or more of the following;

   * Those who have been at least 16 weeks (112 days) and less than 48 weeks (336 days) without additional COVID-19 vaccination since the last COVID-19 vaccination.
   * Those who have been at least 16 weeks (112 days) or more and less than 48 weeks (336 days) since the release of quarantine due to COVID-19 confirmation.
3. Individual with body mass index (BMI) of 30.0 kg/m2 or less at screening visit.
4. Individual who agrees with using an effective birth control method for at least 4 weeks before the screening and during the study period.
5. Individual who agrees not to donate or transfuse blood (including whole blood, plasma components, platelet components, and platelet plasma components) during the study period.

Exclusion Criteria:

1. Individual who has history of COVID-19 or is considered infected within 16 weeks (112 days) prior to administration of investigational product.
2. Individual who has received other COVID-19 vaccine within 16 weeks (112 days) prior to administration of investigational product.
3. Individual who has been in close contact with a COVID-19 infected person, or has been classified as a confirmed or suspected COVID-19 patient within 14 days prior to administration of investigational product.
4. Individual determined to be clinically significantly abnormal by the screening outcome based on laboratory evaluations, electrocardiogram (ECG) and Chest X-ray.
5. Individual who has ant results of positive to HIV test, hepatitis B test, and hepatitis C test on screening.
6. Acute febrile illness with 38°C and above, or any suspected infectious diseases, or symptoms similar to COVID-19 (cough, shortness of breathe, chills, myalgia, headache, sore throat, loss of taste/smell, etc.) within 3 days prior to administration of investigational product.
7. Any serious medical or psychiatric disease which in opinion of investigator judges unable to participate

   * Respiratory diseases: Asthma, Chronic Obstructive Lung Disease (COPD), active or latent tuberculosis which require medication, or individual who has received treatment due to worsening of the respiratory disease within 5 years prior to administration of investigational product.
   * Serious cardiovascular diseases: Congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, myocarditis, pericarditis, etc.
   * Neurologic diseases: Epilepsy, seizure within 3 years, migraine, stroke, encephalopathy, Guillain-Barre Syndrome, encephalomyelitis, acute transverse myelitis, etc.
   * Malignant cancer diagnosed within the past 5 years (skin basal cell and squamous cell carcinoma are excluded).
   * Immune function disorders including autoimmune hypothyroidism, psoriasis.
   * Auto-immune diseases.
   * History of dependently administering psychotropic drugs or narcotic painkillers within 24 weeks prior to administration of investigational product, or psychiatric disease or behavioral impairment that, in the opinion of the investigator, could interfere with the participant's ability to participate in the trial.
   * Other hepatobiliary, renal, endocrine, urinary tract, muscular skeletal diseases which the investigator considers clinically significant.
8. History of splenectomy.
9. History of SARS-CoV or MERS-CoV infection.
10. Known history of allergic or hypersensitivity to the components of investigational product.
11. Known history of serious adverse reactions, allergies or hypersensitivity related to vaccination.
12. History of urticaria within 5 years prior to administration of investigational product.
13. Individual with history of bleeding diathesis or thrombocytopenia, or history of severe bleeding or bruising after intramuscular or intravenous injection, or is receiving an anticoagulant (Those who receive low dose aspirin (less than 100mg/day) are not excluded).
14. Individual with hereditary or idiopathic angioneurotic edema.
15. Individual with solid organ or bone marrow transplantation.
16. Individual who is suspected or with history of substance abuse and alcohol abuse within 24 weeks prior to administration of investigational product.
17. History of SARS-CoV or MERS-CoV vaccination.
18. History of licensed drug for COVID-19 treatment or prevention aside from COVID-19 vaccine within 52 weeks prior to administration of investigational product.
19. Use of immunosuppressive or chronic use of systemic steroids within 6 weeks prior to administration of investigational product (External steroids, nasal spray and inhalants are allowed).

    * Immunosuppressive: Azathioprine, Cyclosporine, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, Cyclophosphamide, 6-Mercaptopurine, Methotrexate, Rapamycin, Leflunomide, etc.
    * Chronic steroid: >10 mg/day prednisone equivalent for periods exceeding 14 days)
20. Individuals who has administered other investigational product or device within 24 weeks prior to screening visit.
21. Individual concomitantly enrolled or scheduled to be enrolled in another trial (including follow-up period).
22. Individual vaccinated or planned vaccination within 28 days prior and after the administration of investigational product.
23. Receipt of immunoglobulin or blood-derived products within 12 weeks prior to administration of investigational product.
24. Individual with scheduled surgery during the study period.
25. Pregnant or lactating women.
26. Individual directly related to the investigator and meets the following conditions:

    * Personnel relationship or subordinate-superior relationship (employees of the investigator's department, staffs of this trial)
    * Students or researchers in the immediate department of the school to which the investigator belongs (e.g., medical university)
27. Individual who is unfit for this study for any other reason in judgement of investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of immediate adverse events (AE) | Within 30 minutes post dose injection
  Proportion of immediate AE within 30 minutes post dose injection.
Proportion of solicited local and systemic AE | Within 7 days (Days 0 - 6) post dose injection
  Proportion of solicited local and systemic AEs within 7 days post dose injection. Local AEs at the site of injection: Pain, tenderness, erythema/redness, swelling/induration, pruritis. Systemic AEs: Fever, fatigue/general weakness, chill, headache, myalgia, arthralgia, diarrhea, nausea/vomiting, abdominal pain, mucocutaneous reaction/rash, urticaria, dizziness, cough, dyspnea.
Proportion of unsolicited AE | Within 28 days post dose injection
  Proportion of unsolicited AEs within 28 days post dose injection. Unsolicited AEs are all other adverse events (those that do not fall under the categories of solicited AEs).
Proportion of SAE | Throughout the study duration, 12 months post dose injection
  Proportion of any SAE from the administration throughout the entire study. An AE or suspected adverse reaction is considered "serious": Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above.
Proportion of Adverse Event Of Special Interest (AESI) | Throughout the study duration, 12 months post dose injection
  Proportion of any AESI from the administration throughout the entire study. AESI are categorized into 1) AESIs included because they are seen with COVID-19 Disease, 2) AESI included because they have a proven or theoretical association with immunization in general, 3) AESI included because they have a proven or theoretical association with specific vaccine platform(s).
Proportion of Medically-Attended Adverse Events (MAAE) | Throughout the study duration, 12 months post dose injection
  Proportion of any MAAE from the administration throughout the entire study. Medically-attended AEs are AEs with medically-attended visits including hospital, emergency room, or other visits to or from medical personnel for any reason. Routine study visits will not be considered medically attended visits.
Proportion of clinically significant changes in clinical safety laboratory parameters | At 7, 14, 28 days post dose injection
  Proportion of clinically significant changes in clinical safety laboratory parameters at 7, 14, 28 days post dose injection.
Proportion of participants achieving seroresponse of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4 weeks post dose injection (Neutralizing antibody) | At 2, 4 weeks post dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 2-fold increase from baseline) of wild-type virus neutralizing antibody titer from baseline to 2, 4 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Geometric Mean Titer of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4 weeks post dose injection (Neutralizing antibody) | At 2, 4 weeks post dose injection
  Geometric Mean Titer (GMT) of neutralizing antibody to the SARS-CoV-2 B.1.1.529 measured by wild-type virus neutralization assay from baseline to 2, 4 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Geometric Mean Fold Rise of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4 weeks post dose injection (Neutralizing antibody) | At 2, 4 weeks post dose injection
  Geometric Mean Fold Rise (GMFR) of neutralizing antibody to the SARS-CoV-2 B.1.1.529 measured by wild-type virus neutralization assay from baseline to 2, 4 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.

SECONDARY OUTCOMES:
Proportion of participants achieving seroresponse of 1 dose of AdCLD-CoV19-1 OMI from baseline to 12, 26, 52 weeks post dose injection (Neutralizing antibody) | At 12, 26, 52 weeks post dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 2-fold increase from baseline) of wild-type virus neutralizing antibody titer from baseline to 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Geometric Mean Titer of 1 dose of AdCLD-CoV19-1 OMI from baseline to 12, 26, 52 weeks post dose injection (Neutralizing antibody) | At 12, 26, 52 weeks post dose injection
  Geometric Mean Titer (GMT) of neutralizing antibody to the SARS-CoV-2 B.1.1.529 measured by wild-type virus neutralization assay from baseline to 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Geometric Mean Fold Rise of 1 dose of AdCLD-CoV19-1 OMI from baseline to 12, 26, 52 weeks post dose injection (Neutralizing antibody) | At 12, 26, 52 weeks post dose injection
  Geometric Mean Fold Rise (GMFR) of neutralizing antibody to the SARS-CoV-2 B.1.1.529 measured by wild-type virus neutralization assay from baseline to 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Proportion of participants achieving seroresponse of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4, 12, 26, 52 weeks post dose injection (ELISA) | At 2, 4, 12, 26, 52 weeks post dose injection
  Proportion of participants achieving seroresponse (SR defined as at least 2-fold increase from baseline) of SARS-CoV-2 B.1.1.529 Spike-binding ELISA IgG antibody from baseline to 2, 4, 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
GMT of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4, 12, 26, 52 weeks post dose injection (ELISA) | At 2, 4, 12, 26, 52 weeks post dose injection
  GMT of SARS-CoV-2 B.1.1.529 Spike-binding ELISA IgG antibody from baseline to 2, 4, 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
GMFR of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4, 12, 26, 52 weeks post dose injection (ELISA) | At 2, 4, 12, 26, 52 weeks post dose injection
  GMFR of SARS-CoV-2 B.1.1.529 Spike-binding ELISA IgG antibody from baseline to 2, 4, 12, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Cell Mediated Immunity (CMI) of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 26, 52 weeks post dose injection (Proportion of responders by Interferon-γ (IFN-γ) ELISpot) | At 2, 26, 52 weeks post dose injection
  Proportion of responders as measured by Interferon-γ (IFN-γ) ELISpot from baseline to 2, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
Cell Mediated Immunity (CMI) of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 26, 52 weeks post dose injection (Median spot forming units by Interferon-γ (IFN-γ) ELISpot) | At 2, 26, 52 weeks post dose injection
  Median spot forming units as measured by Interferon-γ (IFN-γ) ELISpot from baseline to 2, 26, 52 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.

OTHER OUTCOMES:
SRR, GMT, GMFR of 1 dose of AdCLD-CoV19-1 OMI from baseline to 4 weeks post dose injection (Neutralizing antibody) | At 4 weeks post dose injection
  SRR, GMT, GMFR of neutralizing antibody to the SARS-CoV-2 Wuhan strain and Variants of concern (VOC) measured by wild-type virus neutralization assay from baseline to 4 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI.
SRR, GMT, GMFR of 1 dose of AdCLD-CoV19-1 OMI from baseline to 2, 4 weeks post dose injection (Neutralizing antibody) according to the recipients features. | At 2, 4 weeks post dose injection
  SRR, GMT, GMFR of neutralizing antibody to the SARS-CoV-2 B.1.1.529 measured by wild-type virus neutralization assay from baseline to 2, 4 weeks post dose injection induced by 1 dose of AdCLD-CoV19-1 OMI according to the recipients features as follows;
  * Types of last administered COVID-19 vaccines.
  * COVID-19 vaccination order
  * History of COVID-19 infection
  * SARS-CoV-2 N protein status (positive or negative)
Number of virologically-confirmed COVID-19 cases from 2 weeks post dose injection to the end of study period | Throughout the study duration, 12 months post dose injection
  Number of virologically-confirmed COVID-19 cases using Rapid Antigen Test Kit or RT-PCR from 2 weeks post dose injection to the end of study period with one or more symptoms of COVID-19 including fever, chill, cough, shortness of breath, fatigue, myalgia, headache, loss of taste or smell, pharyngitis, rhinorrhea, nausea, vomiting, diarrhea.
Number of severe COVID-19 cases from 2 weeks post dose injection to the end of study period | Throughout the study duration, 12 months post dose injection
  Number of severe COVID-19 cases using Rapid Antigen Test Kit or RT-PCR from 2 weeks post dose injection to the end of study period with one or more symptoms of COVID-19 including:
  * Clinical signs indicative of severe systemic illness (respiratory rate ≥30 per minute, heart rate ≥125 beats per minute, SpO2 ≤93% on room air at sea level or PaO2/FIO2<300 mmHg)
  * Respiratory failure or ARDS (defined as needing high-flow oxygen, non-invasive or mechanical ventilation, or ECMO)
  * Evidence of shock (systolic blood pressure <90 mmHg, diastolic BP <60 mmHg or requiring vasopressors)
  * Significant acute renal, hepatic, or neurologic dysfunction
  * Admission to an intensive care unit or death
Number of hospitalization due to COVID-19 from 2 weeks post dose injection to the end of study period | Throughout the study duration, 12 months post dose injection
  Number of hospitalization due to COVID-19 confirmed by using Rapid Antigen Test Kit or RT-PCR from 2 weeks post dose injection to the end of study period.
Number of death due to COVID-19 from 2 weeks post dose injection to the end of study period | Throughout the study duration, 12 months post dose injection
  Number of death due to COVID-19 confirmed by using Rapid Antigen Test Kit or RT-PCR from 2 weeks post dose injection to the end of study period.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - The Catholic University of Korea ST. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No